CLINICAL TRIAL: NCT02342093
Title: Effects of Two Contraceptives Containing Drospirenone on Blood Pressure in Normotensive Women: a Randomized Controlled Trial
Brief Title: Contraceptives Containing Drospirenone and Blood Pressure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Carolina Sales Vieira, Professor of Obstetrics and Gynecology, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: USP-DRSP
Record Dates: First submitted 2015-01-14; First posted 2015-01-19 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Blood Pressure; Contraception
Keywords: Ambulatory Blood Pressure Monitoring; Drospirenone; Oral contraceptive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 30EE+DRSP (Active Comparator): Combined oral contraceptive containing 30 mcg of ethinylestradiol + 3 mg of drospirenone (30EE+DRSP), 1 pill once a day with a pause of seven days between the blisters for 6 months
  Interventions: Drug: 30EE+DRSP
- 20EE+DRSP (Active Comparator): Combined oral contraceptive containing 20 mcg of ethinylestradiol + 3 mg of drospirenone (20EE+DRSP), 1 pill once a day with a pause of four days between the blisters for 6 months
  Interventions: Drug: 20EE+DRSP

INTERVENTIONS:
Drug: 30EE+DRSP — Combined oral contraceptive containing 30 mcg of ethinylestradiol + 3 mg of drospirenone (30EE+DRSP), 1 pill once a day with a pause of seven days between the blisters for 6 months
  Arms: 30EE+DRSP
Drug: 20EE+DRSP — Combined oral contraceptive containing 30 mcg of ethinylestradiol + 3 mg of drospirenone (20EE+DRSP), 1 pill once a day with a pause of four days between the blisters for 6 months
  Arms: 20EE+DRSP

SUMMARY:
Background: Drospirenone (DRSP) seems to have a favorable effect on blood pressure (BP); however, when associated with ethinylestradiol (EE), this effect does not seem to occur. This study has the objective to assess possible differences in BP associated with the use of COCs containing DRSP with different doses of ethinylestradiol.

Materials and methods: This open-label parallel-group randomized clinical trial involved women randomized to use either 30 mcg of EE+DRSP (n=22) or 20 mcg of EE+DRSP (n=22). Daytime, nighttime and 24-hour BP were evaluated by ambulatory blood pressure monitoring (ABPM) at the beginning of the trial and six months after drug therapy.

ELIGIBILITY:
Inclusion Criteria:

* sexually active women who did not wish to become pregnant,
* aged between 18 and 35,
* with menstrual cycles lasting between 24 and 32 days,
* body mass index (BMI) between 18.0 and 29.9 kg/m2

Exclusion Criteria:

* smoking,
* use of drugs and/or alcohol,
* clinical and/or laboratory signs of hyperandrogenism,
* use of hormonal contraception within six months before the initiation of the study,
* presence of chronic and/or acute inflammatory processes,
* use of medications with endothelial effects (e.g., statins),
* breastfeeding or having stopped breastfeeding within two months before the initiation of the study,
* medical conditions classified as category 3 or 4 according to the WHO medical eligibility criteria for contraceptive prescription

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2011-01; Primary Completion 2013-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 24 hours
  Twenty-four-hour mean systolic blood pressure (SBP), 24-hour mean diastolic blood pressure (DBP), and day and nighttime SBP and DBP were measured by ambulatory blood pressure monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Carolina S Vieira, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil